CLINICAL TRIAL: NCT00211991
Title: A Phase 3, Multicenter, Double-Blinded, Randomized, Study to Compare Immunogenicity and Safety Between Three Commercial Lots of StaphVAX®, a Bivalent Staphylococcus Aureus Glycoconjugate Vaccine in Normal, Healthy, Adult Volunteers
Brief Title: Evaluation of Consistency of StaphVAX Manufacturing Lots
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nabi Biopharmaceuticals (Industry)
Collaborators: Vanderbilt University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Nabi-1369
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2012-05-14 (Estimated); Status verified 2012-05

CONDITIONS: Staphylococcal Infections
MeSH Terms: conditions — Staphylococcal Infections

INTERVENTIONS:
Biological: S. aureus Type 5 & 8 Capsular Polysaccharide Conjugate

SUMMARY:
This study answers a U.S. Food and Drug Administration requirement for evaluation in people of the consistency of manufacturing of a vaccine. Subjects are randomized to one of three lots of vaccine. The antibodies in the blood measure the immunogenicity of each lot of vaccine, and typical vaccine safety information is also collected.

ELIGIBILITY:
Inclusion Criteria:

* healthy,
* written informed consent,
* negative serum pregnancy test if appropriate,
* expect to comply with protocol procedures and schedule

Exclusion Criteria:

* known HIV,
* immunomodulatory drugs,
* malignancy (other than basal cell or squamous cell carcinoma, carcinoma in situ of the cervix, or early stage prostate cancer),
* active infection in the 2 weeks prior to study injection,
* serious S. aureus infection within the last 3 months prior to injection,
* use of investigational drugs, vaccines or devices within the prior 30 days,
* hypersensitivity to components of StaphVAX

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 354
Dates: Start 2005-04; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Type-specific antibody concentrations 6 weeks after vaccine dose.

SECONDARY OUTCOMES:
Antibody concentrations at other time points.
Elicited health events.

CONTACTS AND LOCATIONS:
Overall Officials: Matt Hohenboken, MD, PhD, Study Director — Nabi Biopharmaceuticals
Locations (1):
- Vanderbuilt University, Nashville, Tennessee, United States

REFERENCES:
- [Derived] Creech CB 2nd, Johnson BG, Alsentzer AR, Hohenboken M, Edwards KM, Talbot TR 3rd. Vaccination as infection control: a pilot study to determine the impact of Staphylococcus aureus vaccination on nasal carriage. Vaccine. 2009 Dec 10;28(1):256-60. doi: 10.1016/j.vaccine.2009.09.088. Epub 2009 Sep 30. PMID 19799842